CLINICAL TRIAL: NCT02717897
Title: Association Between Vitamin D Level and Disease Activity in Ulcerative Colitis
Brief Title: Vitamin D and Disease Activity in Ulcerative Colitis
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 11-0202
Record Dates: First submitted 2016-03-10; First posted 2016-03-24 (Estimated); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — 1. Serum
  2. Colon mucosal RNA
  3. Formalin fixed paraffin embedded colon biopsy
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No intervention — This study is not interventional

SUMMARY:
The purpose of this study is to test blood and tissue samples of people with Ulcerative Colitis (UC) to see what effects vitamin D may have on the immune system. This research is being done because it could lead to the development of new treatment for people with inflammatory Bowel Disease (IBD).

DETAILED DESCRIPTION:
Patients with UC will be recruited and consented prior to colonoscopy or flexible sigmoidoscopy. All patients will be age 18 or older with a known history of UC that has been confirmed by biopsy and an extent of disease of at least 20cm proximal to the anus. Clinical data will be collected on the patient's age, disease duration, family history of IBD, smoking status and history, as well as current medications for IBD through a questionnaire. Data will also be collected regarding current vitamin D supplementation (if taking) and dose. Prior to the endoscopic procedure, peripheral blood will be drawn into two 10ml red top tubes. At the time of endoscopy, five standard size mucosal pinch biopsies will be obtained from 20cm proximal to the anus. . A bar-coded unique identifier label will be applied to each sample. One biopsy will be placed in formalin. Paraffin samples will be maintained at room temperature. Following to the endoscopic procedure, the patient's physician will complete a Mayo score based on the patients current symptoms and endoscopic disease severity. Comparison will be made between disease activity, serum serum 25 hydroxyvitamin D level, and mucosal expression of tight junction proteins as well as proinflammatory cytokines.

ELIGIBILITY:
Inclusion:

* Age 18 years old and over
* A diagnosis of ulcerative colitis that has been confirmed by biopsy and an extent of disease of at least 20cm proximal to the anus.

Exclusion:

* Age <18 years old
* Diagnosis of Crohn's disease
* Diagnosis of ulcerative colitis with disease extent <20cm proximal to the anus

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Both female and male participants are being studied
Sampling Method: Probability Sample
Enrollment: 248 (Actual)
Dates: Start 2011-11; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
25(OH) Vitamin D level (ng/ml) | 1 day

SECONDARY OUTCOMES:
Mayo Endoscopy Score | 1 day
mucosal zo-1 expression by real time PCR | 1 day
mucosal occludin expression by real time PCR | 1 day
mucosal VDR expression by real time PCR | 1 day
mucosal claudin-2 expression by real time PCR | 1 day
mucosal TNFa expression by real time PCR | 1 day
mucosal IL-8 expression by real time PCR | 1 day
mucosal VDR expression by immunohistochemistry | 1 day
mucosal zo-1 expression by immunohistochemistry | 1 day
mucosal occludin expression by immunohistochemistry | 1 day
mucosal claudin-2 by immunohistochemistry | 1 day

IPD SHARING:
Plan to Share IPD: No